CLINICAL TRIAL: NCT07314931
Title: The Effects of Neuromuscular Training on Knee Biomechanics During Jump-Landing Among College Basketball Players Post ACL Reconstruction and Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Associate Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: USM/JEPeM/KK/25030307
Record Dates: First submitted 2025-12-15; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation; Knee Injuries; Biomechanical Data; Athletic Performance; Physical Fitness; Neuromuscular Training; Basketball Players
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups. The experimental group will complete neuromuscular training (NMT) in addition to their regular basketball training, while the control group will continue with regular basketball training only. Both groups will follow the 12-week program at the same time, and their results will be compared to see whether NMT improves knee movement, stability, and sport performance after ACL reconstruction.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is an open-label study; both participants and investigators are aware of the intervention being administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (NMT) plus Standard Basketball Training (Experimental): Participants in this arm will receive a 12-week neuromuscular training (NMT) program in addition to their regular basketball training. The NMT program will include balance tasks, jump-landing drills, agility exercises, and core strengthening. Sessions will be conducted in parallel with standard basketball practice.
  Interventions: Behavioral: Neuromuscular Training (NMT)
- Standard Basketball Training (No Intervention): Participants in this arm will continue their usual basketball training program for 12 weeks without additional neuromuscular training. Training content and schedule will follow standard team practice routines. This arm will serve as a comparator to evaluate the added effect of NMT.

INTERVENTIONS:
Behavioral: Neuromuscular Training (NMT) — The neuromuscular training (NMT) program is a 12-week behavioral intervention performed 2-3 times per week in addition to regular basketball training. It includes balance tasks, jump-landing drills, agility exercises, and core strengthening to improve knee stability and movement control after ACL reconstruction
  Arms: Neuromuscular Training (NMT) plus Standard Basketball Training

SUMMARY:
Basketball players often injure the anterior cruciate ligament (ACL), a key structure that stabilizes the knee. Even after surgery and standard rehabilitation, many athletes continue to have problems with knee stability, movement control, and performance during jumping and landing. These issues increase the risk of re-injury and can limit their ability to return to competition.

Neuromuscular training (NMT) is a type of exercise program that focuses on improving balance, muscle coordination, and movement patterns. It uses activities such as jump-landing drills, balance tasks, agility exercises, and core training. Previous research shows that NMT can help athletes land more safely, reduce harmful knee movements, and improve sport performance. However, little is known about its long-term benefits in college basketball players who are more than one year post-ACL surgery.

This study aims to evaluate whether a 12-week NMT program, added to standard basketball training, can improve knee biomechanics, stability, and performance in college basketball players with a history of ACL reconstruction. Thirty participants will be randomly assigned to either an NMT group or a control group. Both groups will complete basketball training, but only the NMT group will receive the additional neuromuscular exercises.

Knee movement will be measured using 3D motion capture and force plates, and performance will be tested through vertical jumps and other sport-specific tasks. The main outcomes will include knee angles during landing, ground reaction forces, dynamic stability, and jump height.

The expected outcome is that athletes who undergo NMT will demonstrate safer landing strategies, better knee control, and improved performance compared to those who only receive standard basketball training. These findings may help coaches and healthcare providers design safer, more effective rehabilitation programs for athletes after ACL surgery.

ELIGIBILITY:
Inclusion Criteria:Male college basketball players

Age 18-25 years

History of anterior cruciate ligament (ACL) reconstruction surgery at least 12 months before enrollment

Cleared by physician for sports participation

Willing to provide informed consent and comply with study procedures

Exclusion Criteria:Previous ACL injury on the contralateral knee

Other major lower-limb injuries (e.g., meniscus, cartilage, fractures) in the past 12 months

Current knee pain, swelling, or instability that prevents safe participation

Neurological, cardiovascular, or systemic conditions that may affect training safety

Participation in another structured neuromuscular training program within the past 6 months

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only male college basketball players aged 18-25 years, at least 1 year post-ACL reconstruction, are eligible to participate.
Enrollment: 30 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Peak knee valgus angle during single-leg jump-landing (degrees) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Knee valgus angle will be measured using 3D motion capture during a standardized single-leg jump-landing task. The primary endpoint is the peak knee valgus angle (°) during the landing phase, averaged across 3 successful trials.

SECONDARY OUTCOMES:
Time to stabilization after landing (seconds) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Dynamic postural stability will be evaluated using force platform data during a standardized single-leg jump-landing task. The endpoint is time to stabilization (TTS, s) following landing, averaged across 3 successful trials.
Center of pressure displacement after landing, medial-lateral (millimeters) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Center of pressure (COP) displacement will be quantified from force platform data during a standardized single-leg jump-landing task. The endpoint is COP displacement in the medial-lateral direction (mm), averaged across 3 successful trials.
Peak knee flexion angle during single-leg jump-landing (degrees) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Peak knee flexion angle during the landing phase will be measured using 3D motion capture during a standardized single-leg jump-landing task. The endpoint is the peak knee flexion angle (°), averaged across 3 successful trials.
Center of pressure displacement after landing, anterior-posterior (millimeters) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Center of pressure (COP) displacement will be quantified from force platform data during a standardized single-leg jump-landing task. The endpoint is COP displacement in the anterior-posterior direction (mm), averaged across 3 successful trials.
Countermovement jump height (centimeters) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Explosive lower-limb power will be assessed using a countermovement jump (CMJ) on a force platform. The endpoint is jump height (cm) calculated from flight time, averaged across 3 successful trials.
Squat jump height (centimeters) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Explosive lower-limb power will be assessed using a squat jump (SJ) on a force platform. The endpoint is jump height (cm) calculated from flight time, averaged across 3 successful trials.
Knee flexion angle at initial contact during single-leg jump-landing (degrees) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Knee flexion angle at initial ground contact will be measured using 3D motion capture during a standardized single-leg jump-landing task. The endpoint is the knee flexion angle at initial contact (°), averaged across 3 successful trials.
Peak vertical ground reaction force during single-leg jump-landing (Newtons) | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Vertical ground reaction force (vGRF) will be measured using force platforms during a standardized single-leg jump-landing task. The endpoint is peak vGRF (N) during landing, averaged across 3 successful trials.

OTHER OUTCOMES:
Percentage of prescribed neuromuscular training (NMT) sessions completed | Throughout the 12-week intervention period
  Adherence will be assessed as the percentage of prescribed NMT sessions completed over the 12-week intervention period. A session will be considered completed if the participant attends and completes the full planned session.
Number of participants with ≥1 intervention-related adverse event | Throughout the 12-week intervention period
  Safety will be assessed as the number of participants with ≥1 intervention-related adverse event during the 12-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Chengde Medical University, Affiliated Hospital, Chengde, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR